CLINICAL TRIAL: NCT00336024
Title: A Phase III Randomized Trial for the Treatment of Newly Diagnosed Supratentorial PNET and High Risk Medulloblastoma in Children < 36 Months Old With Intensive Induction Chemotherapy With Methotrexate Followed by Consolidation With Stem Cell Rescue vs. the Same Therapy Without Methotrexate
Brief Title: Combination Chemotherapy Followed By Peripheral Stem Cell Transplant in Treating Young Patients With Newly Diagnosed Supratentorial Primitive Neuroectodermal Tumors or High-Risk Medulloblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0334; NCI-2009-00338 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000483683; 07-654; ACNS0334; COG-ACNS0334; ACNS0334 (Other: Children's Oncology Group); ACNS0334 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anaplastic Medulloblastoma; Medulloblastoma; Supratentorial Embryonal Tumor, Not Otherwise Specified; Untreated Childhood Supratentorial Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Medulloblastoma | interventions — Stem Cell Transplantation; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin; Methotrexate; merphos; Thiotepa; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (induction+consolidation chemotherapy, autologous PBSC) (Active Comparator): Patients receive vincristine IV over 1 minute on days 1, 8, and 15; etoposide IV over 1 hour on days 1-3; cyclophosphamide IV over 1 hour on days 1 and 2; cisplatin IV over 6 hours on day 3. Treatment repeats every 3 weeks for 3 courses.
  Within 6 weeks after completion of induction therapy, patients receive consolidation therapy comprising carboplatin IV over 2 hours and thiotepa IV over 2 hours on days 1 and 2 and G-CSF IV or SC beginning on day 5 and continuing until blood counts recover. Patients also receive autologous PBSC IV on day 4. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Thiotepa; Drug: Vincristine Sulfate
- Arm II (induction+consolidation chemotherapy, autologous PBSC) (Experimental): Patients receive vincristine IV over 1 minute on days 1, 8, and 15; high-dose methotrexate IV over 4 hours on day 1; and leucovorin calcium IV or PO every 6 hours beginning on day 2 and continuing until methotrexate levels are in a safe range. Patients then receive etoposide IV over 1 hour on approximately days 4, 5, and 6, cyclophosphamide IV over 1 hour on approximately days 4 and 5, and cisplatin IV over 6 hours on approximately day 6. Treatment repeats every 3 weeks for 3 courses.
  Within 6 weeks after completion of induction therapy, patients receive consolidation therapy comprising carboplatin IV over 2 hours and thiotepa IV over 2 hours on days 1 and 2 and G-CSF IV or SC beginning on day 5 and continuing until blood counts recover. Patients also receive autologous PBSC IV on day 4. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Methotrexate; Other: Quality-of-Life Assessment; Drug: Thiotepa; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSC resuce
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given IV or SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV or orally
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm II (induction+consolidation chemotherapy, autologous PBSC)
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm II (induction+consolidation chemotherapy, autologous PBSC)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial is studying two different combination chemotherapy regimens to compare how well they work in treating young patients with newly diagnosed supratentorial primitive neuroectodermal tumors or high-risk medulloblastoma when given before additional intense chemotherapy followed by peripheral blood stem cell rescue. It is not yet known which combination chemotherapy regimen is more effective when given before a peripheral stem cell transplant in treating supratentorial primitive neuroectodermal tumors or medulloblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if treatment of infants with high risk primitive neuroectodermal tumors (PNET) central nervous system (CNS) tumors with intensive chemotherapy plus high-dose methotrexate and peripheral blood stem cell rescue results in a higher complete response rate then the same regimen without methotrexate.

SECONDARY OBJECTIVES:

I. To determine whether biologic characterization of these tumors will refine therapeutic stratification separating atypical teratoid rhabdoid tumors (AT/RT) from primitive neuroectodermal tumors (PNETs) and possibly identifying other markers of value for stratification within the group of PNETs.

II. To determine if event free survival (EFS) and patterns of failure differ between the methotrexate arm versus the arm without methotrexate.

III. To compare the acute, chronic and late effects of these two very intensive regimens, especially as to the tolerance of the same consolidation regimen following the differing induction regimens.

IV. To compare the gastrointestinal and nutritional toxicities of these intense regimens.

V. To describe and compare the quality of life outcomes and neuropsychological effects of these intense systemic therapies.

OUTLINE: Patients are randomized to 1 of 2 treatment arms

INDUCTION THERAPY:

ARM I: Patients receive vincristine IV over 1 minute on days 1, 8, and 15; etoposide IV over 1 hour on days 1-3; cyclophosphamide IV over 1 hour on days 1 and 2; cisplatin IV over 6 hours on day 3; and filgrastim (G-CSF) IV or subcutaneously (SC) beginning on day 4 and continuing until blood counts recover. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive vincristine IV over 1 minute on days 1, 8, and 15; high-dose methotrexate IV over 4 hours on day 1; and leucovorin calcium IV or orally (PO) every 6 hours beginning on day 2 and continuing until methotrexate levels are in a safe range. Once methotrexate levels are in a safe range, patients then receive etoposide IV over 1 hour on approximately days 4, 5, and 6, cyclophosphamide IV over 1 hour on approximately days 4 and 5, and cisplatin IV over 6 hours on approximately day 6. Patients also receive G-CSF IV or SC beginning 24 hours after the completion of chemotherapy and continuing until blood counts recover. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

In both arms, patients with stable disease or partial response after induction therapy proceed to second-look surgery followed by consolidation therapy. Patients with a complete response after induction therapy proceed directly to consolidation therapy.

CONSOLIDATION THERAPY: Beginning no more than 6 weeks after completion of induction therapy, patients receive consolidation therapy comprising carboplatin IV over 2 hours and thiotepa IV over 2 hours on days 1 and 2 and G-CSF IV or SC beginning on day 5 and continuing until blood counts recover. Patients also receive autologous peripheral blood stem cells (PBSC) IV on day 4. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically for 4 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* High-risk medulloblastoma defined by any of the following:

  * > 1.5 cm^2 residual disease for any medulloblastoma histology, or
  * Lumbar cerebral spinal fluid (CSF) cytology positive for tumor cells by analysis of fluid collected either before definitive surgery or at least 10 days after definitive surgery unless contraindicated, or
  * Magnetic resonance imaging (MRI) evidence of M2 or M3 metastatic disease, or
  * M4 disease
* Supratentorial primitive neuroectodermal tumor (PNET) (any M-stage) will be eligible for study entry
* Children less than 8 months of age at the time of definitive surgery with or without measurable radiographic residual tumor with M0 stage medulloblastoma will be eligible for study entry
* Patients with anaplastic medulloblastoma are eligible regardless of M-stage or residual tumor
* Patients with M0 classic, non-desmoplastic medulloblastoma (R1) with radiographically measurable residual disease < 1.5 cm^2 are eligible
* Cranial MRI (with and without gadolinium) must be done pre-operatively; post-operatively, cranial MRI (with and without gadolinium) must be done, preferably within 48 hours of surgery; entire spinal MRI must be obtained either pre-operatively (with gadolinium) or post-operatively (at least 10 days following surgery) prior to study enrollment (with and without gadolinium); patients with MRI evidence of spinal disease are eligible for this study
* Evaluation of lumbar CSF cytology (cytospin preparation for microscopic evaluation) must be performed either pre-operatively or at least 10 days after definitive surgery unless contraindicated
* Patient must have a life expectancy > 8 weeks
* Patient must have received no prior radiation therapy or chemotherapy other than corticosteroids; corticosteroids are allowable for all patients
* Creatinine clearance or radioisotope glomerular filtration rate >= 60 mL/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age, and
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic pyruvic transaminase (SGPT) (alanine transaminase [ALT]) < 2 x ULN for age
* Shortening fraction >= 27% by echocardiogram, or
* Ejection fraction >= 47% by radionuclide angiogram
* No evidence of dyspnea at rest
* Pulse oximetry > 94% on room air
* Peripheral absolute neutrophil count (ANC) > 1,000/uL
* Platelet count > 100,000/uL (transfusion independent)
* Hemoglobin greater than 8 g/dL (may have received red blood cell [RBC] transfusions allowed)
* Hold trimethoprim/sulfamethoxazole (Bactrim) on the day of high-dose methotrexate (HDMTX) infusion and continue to hold until the methotrexate level is less than 0.1 micromolar (1 x 10-7 M)
* Avoid probenecid, penicillins, cephalosporins, aspirin, proton pump inhibitors and nonsteroidal anti-inflammatory drug (NSAIDS) on the day of methotrexate and continue until the methotrexate level is less than 0.1 micromolar (1 x 10-7 M) as renal excretion of methotrexate is inhibited by these agents
* Avoid IV contrast media, urinary acidifiers, phenytoin, and fosphenytoin on the day of methotrexate and until the methotrexate level is less than 0.1 micromolar (1 x 10-7 M)
* Concurrent use of enzyme inducing anticonvulsants (e.g. phenytoin, phenobarbital, and carbamazepine) should be avoided
* Clinically significant drug interactions have been reported when using vincristine with strong cytochrome P450 (CYP450) family 3 subfamily A member 4 (3A4) inhibitors and inducers; selected strong inhibitors of cytochrome P450 3A4 include azole antifungals, such as fluconazole, voriconazole, itraconazole, ketoconazole, and strong inducers include drugs such as rifampin, phenytoin, phenobarbitol, carbamazepine, and St. John's wort; the use of these drugs should be avoided with vincristine
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2007-10-22 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Mazewski, Principal Investigator — Children's Oncology Group
Locations (145):
- United States (129):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (11):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- San Jorge Children's Hospital, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children less than 36 months with high risk medulloblastoma/PNET were enrolled in the study. The first eligible patient was enrolled on October 22, 2007 and the last patient was enrolled on April 23, 2014.
Pre-assignment Details: This is a Phase 3 randomized trial designed to determine whether or not the addition of high dose Methotrexate will achieve a higher complete response rate.
Groups:
- Arm I (Patients Treated Without Methotrexate (MTX)): Patients receive vincristine sulfate IV on days 1, 8, and 15; etoposide IV over 1 hour on days 1-3; cyclophosphamide IV over 1 hour on days 1 and 2; cisplatin IV over 6 hours on day 3. Treatment repeats every 3 weeks for 3 courses.
  Within 6 weeks after completion of induction therapy, patients receive consolidation therapy comprising carboplatin IV over 2 hours and thiotepa IV over 2 hours on days 1 and 2 and filgrastim (G-CSF) IV or SC beginning on day 54 and continuing until blood counts recover. Patients also receive autologous PBSC IV on day 4. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
- Arm II (Patients Treated With MTX): Patients receive vincristine sulfate IV on days 1, 8, and 15; high-dose methotrexate IV over 4 hours on day 1; and leucovorin calcium IV or orally every 6 hours beginning on day 2 and continuing until methotrexate levels are in a safe range. Patients then receive etoposide IV over 1 hour on approximately days 4, 5, and 6, cyclophosphamide IV over 1 hour on approximately days 4 and 5, and cisplatin IV over 6 hours on approximately day 6. Treatment repeats every 3 weeks for 3 courses.
  Within 6 weeks after completion of induction therapy, patients receive consolidation therapy comprising carboplatin IV over 2 hours and thiotepa IV over 2 hours on days 1 and 2 and filgrastim (G-CSF) IV or SC beginning on day 54 and continuing until blood counts recover. Patients also receive autologous PBSC IV on day 4. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Started | 46 | 45
Completed | 26 | 26
Not Completed | 20 | 19
Not completed — Death | 2 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Failure to fulfill consolidation | 1 | 1
Not completed — Progressive Disease | 4 | 7
Not completed — Ineligible | 7 | 7

BASELINE CHARACTERISTICS:
Population: Only eligible patients are included in the baseline characteristics. Seven patients were excluded in each treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX) | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.97 (0.75) | 1.73 (0.87) | 1.85 (0.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 15
  Not Hispanic or Latino | 33 | 26 | 59
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Have Either a Complete Response (CR) Rate or No Complete Response Rate
Description: At the end of consolidation, the number of evaluable patients treated with intensive chemotherapy with methotrexate who achieved CR or not will be compared to those who achieved CR or not after treated with the same intensive chemotherapy without methotrexate. The CR rates between these two groups will be compared at a significance level of 0.1 using one-sided Chi-square test. Complete Response (CR) requires: CR for target lesions: disappearance of all target lesions, CR for non-target lesions: disappearance of all non-target lesions and no new lesions. No CR is any response not fitting the definition of CR.
Time Frame: At the end of consolidation treatment
Population: Per protocol, only evaluable patients are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 29 | 30
Participants
  Complete response | 13 | 15
  No Complete response | 16 | 15
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); The CR rates between these two groups will be compared at a significance level of 0.1 using one-sided Chi-square test; Test type: Superiority; p = 0.35, Chi-squared

2. Secondary Outcome: Number of Participants With Molecular Sub-types of MB, CNS-PNETs/EBTs Represented in the ACNS0334 Cohort
Description: The number of patients will be reported for this analysis by Molecular Sub-types of MB, CNS-PNETs/EBTs
Time Frame: At baseline
Population: 13 patients without molecular data, because of lack of sufficient materials or poor quality of the data, were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 34 | 30
Participants
  Medulloblastoma, sonic hedgehog subgroup | 5 | 6
  Medulloblastoma, group 3 subgroup | 15 | 10
  Medulloblastoma, group 4 subgroup | 0 | 2
  Embryonal tumor with multilayered rosettes | 9 | 5
  Pineoblastoma | 3 | 6
  Atypical teratoid/rhabdoid tumor | 1 | 0
  High-grade glioma | 1 | 0
  Pleomorphic xanthoastrocytoma | 0 | 1

3. Secondary Outcome: Percentage of Participants With Event Free Survival (EFS)
Description: EFS was defined as time from enrollment to the occurrence of first event (disease progression/relapse, secondary malignancy, death from any cause) or date of last contact for patients who are event-free. The percentage of participants with EFS and 80% confidence interval were provided. The difference in incidence for the two treatment regimens were compared using a one-sided log-rank test with a significance level of 0.1.
Time Frame: Baseline to up to 5 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Number (80% Confidence Interval); unit: percentage of participants with EFS
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
percentage of participants with EFS | 43.6 [33.3 to 53.4] | 52.6 [41.8 to 62.4]
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); The difference in incidence for the two treatment regimens will be compared using a one-sided log-rank test with a significance level 0.1; Test type: Superiority; p = 0.28, Log Rank

4. Secondary Outcome: Patterns of Failure
Description: The patterns of failure for relapse/disease progression will be provided for patients treated with/without methotrexate drug in three categories, namely local, distant, and both local and distant. The number of patients with each type of failure will be listed per arm. The two groups will be compared to determine if the pattern of failure distribution is different between the two arms using Fisher exact test.
Time Frame: Baseline to up to 5 years
Population: All Eligible Participants who relapsed/disease progressed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 20 | 16
Participants
  Local | 7 | 6
  Distant | 8 | 7
  Both Local and Distant | 5 | 3
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); The two groups will be compared for patterns of failure to detect a statistically significant difference using Fisher exact test; Test type: Superiority; p = 1.00, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Any Acute Adverse Events
Description: Event is defined as the first occurrence of any acute toxicity. Estimates will be obtained using life-table methods. Patients who have progression or recurrence of disease will be censored in this analysis. Difference in incidence for the two treatment regimens will be compared using log-rank test.
Time Frame: Beginning of treatment to the end of consolidation
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
percentage of participants | 97.4 [88.5 to 99.8] | 97.2 [87.7 to 99.8]
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Difference in incidence for the two treatment regimens will be compared using log-rank test; Test type: Superiority; p = 0.74, Log Rank

6. Secondary Outcome: Number of Participants With Acute Hearing Loss and No Acute Hearing Loss
Description: Per protocol, hearing was assessed pretreatment and at regular specified intervals during treatment and off therapy, using DPOAE, audiogram or Brainstem Evoked Auditory. Per CTCAE V4.0 grade 3 Hearing impaired is defined as follows; Pediatric (on a 1,2,3,4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids, threshold shift >20 dB at 3 kHz and above in at least one ear, additional speech-language related services as indicated. Per CTCAE V4.0 grade 4 Hearing impaired is defined as follows; Pediatric Audiologic indication for cochlear implant and additional speech-language related services as indicated.
Time Frame: Beginning of treatment to the end of consolidation
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants
  Acute Hearing Loss | 7 | 6
  No Acute Hearing Loss | 32 | 32
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); The rate of acute hearing loss between two treatment regimens will be be compared using Fisher exact test; Test type: Superiority; p = 1.00, Fisher Exact

7. Secondary Outcome: Number of Participants With Chronic Primary Hypothyroidism/Subclinical Compensatory HypothyroidismHypothyroidism/Subclinical Compensatory Hypothyroidism
Description: Thyroid function was assessed as per ACNS0334 Endocrine Guidelines. "Normal" and "Abnormal" are defined at each institution by the laboratory standards where the blood tests are run. Primary Hypothyroidism/Subclinical Compensatory Hypothyroidism is defined as patients with Free T4 level less than "Institutional" Normal or equal to "Institutional" Normal with TSH level greater than "Institutional" Normal.
Time Frame: Off-treatment up to 9 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants | 3 | 5

8. Secondary Outcome: Number of Participants With Chronic Central Hypothyroidism
Description: Thyroid function was assessed as per ACNS0334 Endocrine Guidelines. "Normal" and "Abnormal" are defined at each institution by the laboratory standards where the blood tests are run. Central Hypothyroidism is defined as Free T4 level less than "Institutional" Normal with TSH less than or equal to "Institutional" Normal.
Time Frame: Off-treatment up to 9 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants | 1 | 1

9. Secondary Outcome: Number of Participants With Chronic Low Somatomedin C
Description: Low Somatomedin C is defined as patients with somatomedin C value less than institutional normal. As numbers are too small, descriptive statistics such as number will be reported for this analysis. Growth hormone function was assessed as per ACNS0334 Endocrine Guidelines. Low Somatomedin C levels are defined at each institution by the laboratory standards where the blood tests are run.
Time Frame: Off-treatment up to 9 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants | 2 | 5

10. Secondary Outcome: Number of Participants With Chronic Diabetes Insipidus
Description: The number of patients who had "Diabetes Insipidus" and on DDAVP will be reported for this analysis due to small numbers..
Time Frame: Beginning of off-treatment to up to 9 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants | 1 | 1

11. Secondary Outcome: Number of Participants With Secondary Malignancies
Description: The number of patients who had secondary malignancy will be reported for this analysis due to small numbers.
Time Frame: Off-treatment up to 9 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants | 1 | 0

12. Secondary Outcome: Number of Participants With Chronic/Late Hearing Loss and No Chronic/Late Hearing Loss
Description: The number of patients who are reported to have abnormal hearing, graded according to CTCAE 4.0 or not, with onset while on therapy or when off therapy which persisted after off therapy will be reported and will be compared using Fisher exact test.
Time Frame: Off-treatment up to 9 years
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants
  Chronic/Late Hearing Loss | 12 | 13
  No Chronic/Late Hearing Loss | 27 | 25
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); The rate of chronic hearing loss between two treatment regimens will be be compared using Fisher exact test; Test type: Superiority; p = 0.8, Fisher Exact

13. Secondary Outcome: Rates of Gastrointestinal Toxicities
Description: Rates of gastrointestinal toxicities reported as Adverse Events during therapy for each cycle will be summarized using standard descriptive methods (such as number of patients). The difference in number of patients with gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test.
Time Frame: Beginning of treatment to the end of consolidation
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants
  GI Tox Induction Cycle I | 8 | 12
  No GI Tox Induction Cycle I | 31 | 26
  GI Tox Induction Cycle II | 4 | 10
  No GI Tox Induction Cycle II | 35 | 28
  GI Tox Induction Cycle III | 4 | 8
  No GI Tox Induction Cycle III | 35 | 30
  GI Tox Consolidation Cycle I | 11 | 14
  No GI Tox Consolidation Cycle I | 28 | 24
  GI Tox Consolidation Cycle II | 7 | 10
  No GI Tox Consolidation Phase II | 32 | 28
  GI Tox Consolidation Cycle III | 5 | 6
  No GI Tox Consolidation Cycle III | 34 | 32
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of gastrointestinal toxicities in Induction Phase I. The difference in number of patients with/without gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.27, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of gastrointestinal toxicities in Induction Phase II. The difference in number of patients with/without gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.07, Chi-squared
Statistical Analysis 3: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of gastrointestinal toxicities in Induction Phase III. The difference in number of patients with/without gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.2, Chi-squared
Statistical Analysis 4: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of gastrointestinal toxicities in Consolidation Phase 1. The difference in number of patients with/without gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.4, Chi-squared
Statistical Analysis 5: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of gastrointestinal toxicities in Consolidation Phase 2. The difference in the number of patients with/without gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.38, Chi-squared
Statistical Analysis 6: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of gastrointestinal toxicities in Consolidation Phase III. The difference in number of patients with/without gastrointestinal toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.7, Chi-squared

14. Secondary Outcome: Rates of Nutritional Toxicities
Description: Rates of nutritional toxicities reported as Adverse Events during therapy for each cycle will be summarized using standard descriptive methods (such as number of patients). The difference in number of patients with nutritional toxicities between the two treatment regimens will be compared using a Chi-square test.
Time Frame: Beginning of treatment to the end of consolidation
Population: Per protocol all eligible patients randomized to treatment should be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 39 | 38
Participants
  Nutritional Disorders Induction Cycle I | 10 | 17
  No Nutritional Disorders Induction Cycle I | 29 | 21
  Nutritional Disorders Induction Cycle II | 13 | 13
  No Nutritional Disorders Induction Cycle II | 26 | 25
  Nutritional Disorders Induction Cycle III | 7 | 12
  No Nutritional Disorders Induction Cycle III | 32 | 26
  Nutritional Disorders Consolidation Cycle I | 12 | 8
  No Nutritional Disorders Consolidation Cycle I | 27 | 30
  Nutritional Disorders Consolidation Cycle II | 9 | 5
  No Nutritional Disorders Consolidation Cycle II | 30 | 33
  Nutritional Disorders Consolidation Cycle III | 10 | 5
  No Nutritional Disorders Consolidation Cycle III | 29 | 33
Statistical Analysis 1: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of nutritional toxicities in Induction Phase I. The difference in number of patients with/without nutritional toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.08, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of nutritional toxicities in Induction Phase II. The difference in number of patients with/without nutritional toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.9, Chi-squared
Statistical Analysis 3: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of nutritional toxicities in Induction Phase III. The difference in number of patients with/without nutritional toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.17, Chi-squared
Statistical Analysis 4: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of nutritional toxicities in Consolidation Phase I. The difference in number of patients with/without nutritional toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.3, Chi-squared
Statistical Analysis 5: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of nutritional toxicities in Consolidation Phase II. The difference in number of patients with/without nutritional toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.26, Chi-squared
Statistical Analysis 6: Comparison: Arm I (Patients Treated Without Methotrexate (MTX)) vs Arm II (Patients Treated With MTX); Rates of nutritional toxicities in Consolidation Phase III. The difference in number of patients with/without nutritional toxicities between the two treatment regimens will be compared using a Chi-square test; Test type: Superiority; p = 0.17, Chi-squared

15. Secondary Outcome: Median/Range of Patients for Total Quality of Life (QOL) Score, Intelligence Quotient (IQ) and Processing Speed Index (PSI).
Description: Three tools are used to assess intelligence (IQ) depending on age. The range of IQ scores is 40-160 (mean=100, SD=15); range for the Processing Speed Index (PSI)=45-155. Higher scores represent better functioning. (1) Wechsler Preschool and Primary Scale of Intelligence-4th Edition (WPPSI-IV) is used for ages 2.5 to 6 years. Bug Search and Cancellation subtests are summed to calculate PSI. (2) Wechsler Intelligence Scales for Children-5th Edition (WISC-V) is used for ages 6 - 16 years. Symbol Search and Coding subtests are summed to calculate PSI. (3) Wechsler Adult Intelligence Scales-4th Edition (WAIS-IV) is used for ages 16 and older. Symbol Search and Coding subtests are summed to calculate PSI.
  The Pediatric Quality of Life Inventory Version 4 (PedsQL) measures health-related quality of life (QOL). Parents complete the measure for children ages 2-17, and patients > 18 complete a self-report version. Total scores range from 0-100, with higher scores representing better QOL.
Time Frame: 60 months (+/- 3 months)
Population: Of the 77 eligible participants in ACNS0334, only 4 patients completed assessments in ALTE07C1 study. The targeted number of participants to achieve target power and statistically reliable results was not achieved and therefore the data is statistically uninterpretable.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
Number analyzed (Participants) | 2 | 2
scores on a scale
  Total Quality of Life Score | 60.5 [54.0 to 67.0] | 56.5 [35.0 to 78.0]
  Intelligence Quotient | 77.0 [71.0 to 83.0] | 78.5 [74.0 to 83.0]
  Processing Speed Index: number analyzed (Participants) | 2 | 1
  Processing Speed Index | 82.0 [78.0 to 86.0] | 89.0 [89.0 to 89.0]

ADVERSE EVENTS:
Description: Adverse Events/Serious Adverse Events were reported for all eligible patients (n=77) by treatment arm in the study. The total number of participants at risk represents total number of eligible patients in the study by treatment arm.
Arm/Group | Arm I (Patients Treated Without Methotrexate (MTX)) | Arm II (Patients Treated With MTX)
All-Cause Mortality (participants affected / at risk) | 18/39 | 15/38
Serious Adverse Events (participants affected / at risk) | 8/39 | 3/38
Other Adverse Events (participants affected / at risk) | 39/39 | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm I (Patients Treated Without Methotrexate (MTX)) (N=39) | Arm II (Patients Treated With MTX) (N=38)
Colitis (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Death NOS, Related to progressive disease and not due to protocol therapy (General disorders) | 1 (1) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0/0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0/0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
osteosarcoma in field of radiation administered for first recurrence, p53 predisposition syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Patients Treated Without Methotrexate (MTX)) (N=39) | Arm II (Patients Treated With MTX) (N=38)
Anemia (Blood and lymphatic system disorders) | 31 (122) | 19 (84)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (53) | 20 (43)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 7 (12) | 6 (6)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 4 (6) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 11 (12) | 7 (10)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 3 (3)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 5 (6) | 13 (21)
Nausea (Gastrointestinal disorders) | 5 (7) | 3 (5)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 3 (6)
Vomiting (Gastrointestinal disorders) | 11 (13) | 12 (22)
Death NOS (General disorders) | 2 (2) | 3 (3)
Fever (General disorders) | 1 (1) | 4 (5)
Irritability (General disorders) | 1 (1) | 2 (3)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 5 (7)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 6 (6) | 8 (16)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 7 (11)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 22 (47) | 18 (45)
Lung infection (Infections and infestations) | 0 (0) | 2 (3)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 5 (7)
Skin infection (Infections and infestations) | 0 (0) | 3 (3)
Small intestine infection (Infections and infestations) | 0 (0) | 2 (2)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4) | 4 (5)
Wound infection (Infections and infestations) | 0 (0) | 4 (6)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Venous injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (16) | 21 (39)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 12 (20)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 3 (5) | 2 (5)
Lymphocyte count decreased (Investigations) | 18 (63) | 14 (80)
Neutrophil count decreased (Investigations) | 31 (127) | 28 (125)
Platelet count decreased (Investigations) | 32 (150) | 27 (139)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 30 (122) | 22 (118)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (17) | 9 (20)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (7) | 8 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 17 (31) | 17 (30)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 9 (9) | 9 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (12) | 8 (9)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 3 (3) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 5 (9)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 4 (6)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.